CLINICAL TRIAL: NCT05894928
Title: A Phase 1 Study to Investigate the Effect of Cholestyramine on the Pharmacokinetics of LOXO-783 in Healthy Adults
Brief Title: A Study to Evaluate the Effect of Cholestyramine on LOXO-783 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-PIK-23009; J4C-OX-JZUD (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-06; First posted 2023-06-08 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Cholestyramine; LOXO-783
MeSH Terms: interventions — Cholestyramine Resin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LOXO-783 alone (Experimental): Single dose of LOXO-783 administered orally.
  Interventions: Drug: LOXO-783
- LOXO-783 + Cholestyramine 1 hour post dose (Experimental): Single dose of LOXO-783 administered orally followed by a single dose of cholestyramine administered orally after 1 hour.
  Interventions: Drug: LOXO-783; Drug: Cholestyramine
- LOXO-783 + Cholestyramine 4 hours post dose (Experimental): Single dose of LOXO-783 administered orally followed by a single dose of cholestyramine administered orally after 4 hours.
  Interventions: Drug: LOXO-783; Drug: Cholestyramine

INTERVENTIONS:
Drug: LOXO-783 — Administered orally.
  Other Names: LY3849524
Drug: Cholestyramine — Administered orally.
  Arms: LOXO-783 + Cholestyramine 1 hour post dose; LOXO-783 + Cholestyramine 4 hours post dose

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much LOXO-783 is in the bloodstream and how the body handles and eliminates LOXO-783 when administered alone or in combination with cholestyramine in healthy participants. The study will also evaluate the safety and tolerability of LOXO-783 with and without cholestyramine. Participation could last up to 63 days including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status as defined by the absence of evidence of any clinically significant active or chronic disease
* Body mass index (BMI): 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Females who are lactating or of childbearing potential
* Clinically significant history of any drug sensitivity, drug allergy, or food allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LOXO-783 | Predose on Day 1 upto 96 hours postdose of each treatment period
  PK: Cmax of LOXO-783
PK: Area Under the Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC[0-inf]) of LOXO-783 | Predose on Day 1 upto 96 hours postdose of each treatment period
  PK: AUC(0-inf) of LOXO-783

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, MD; PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Labcorp Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No